CLINICAL TRIAL: NCT07039344
Title: Effectiveness of Palliative Care Training Program Among Senior Student Nurses And Its Impact In Experiential Learning In Nursing Education
Brief Title: Effectiveness of Palliative Care Training and Its Impact on Experiential Learning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lincoln University College Malaysia (Other)
Responsible Party: Principal Investigator, Mishal Liaqat, student, Lincoln University College Malaysia
Organization: Lincoln University College (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LUC/CGPS/0614032022
Record Dates: First submitted 2025-05-21; First posted 2025-06-26 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Support, Family; The Effects of Educational Intervention on Nurses Performance
Keywords: Palliative care; palliative care education; compare

STUDY DESIGN:
Intervention Model Description: There will be two groups receiving two different intervention simultaneously. so the best mode match my study is parallel
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants of both groups remained uninformed regarding their allocation status by conducting study at two different nursing colleges. Group A intervention will be provided in Rai foundation College of Nursing, Sargodha. The group B will be provided intervention at Al-Aleem Institute of Nursing, Lahore, Pakistan. So, through geographical space masking of participants will be possible. The facilitators / evaluators, who assessed the student's competency, shall remain uninformed regarding the student's allocation status in the post-assessment to minimize the risk of bias and make the assessment more objective.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional method of Palliative care Training (Group A) (Active Comparator): Group A receive training through the 2-step Conventional method. The first step comprises lectures followed by skill session. The lecture content will be the same for both groups. The students practiced their skills under instructor supervision on the manikins in groups of 5 students in each group. The errors will be corrected on the spot.
  Interventions: Other: Conventional method of Palliative care Training (Group A)
- Pedagogical (LWPPR) method of Palliative care Training (Group B) (Experimental): Group B will receive training through the 5-steps pedagogy method including: the 1st step (learn), in which didactic lectures will be given to the students leading to the 2nd step (video watch), a 30 minutes video on Palliative care. The students first see the video in the class on multimedia with explanation and then share to the students in what's up group for frequent watching as per need. In the 3rd step (practice), students practiced their skills on a low fidelity simulator under instructor supervision on a scheduled day of the week in the nursing skill lab for 6 weeks. The errors will be corrected on the spot. A total of 10 groups will make with a ratio of 10 in each group. In the 4th step (perform), students perform their skill in real-life situations through the clinical rotation under supervision. Finally, the 5th step (Retain) will be established through self-directed learning in which an additional one-hour skill session / week will be provided to the students.
  Interventions: Other: Pedagogical (LWPPR) method of Palliative care Training (Group B)

INTERVENTIONS:
Other: Conventional method of Palliative care Training (Group A) — Group A receive training through the 2-step Conventional method. The first step comprises 1 didactic lecture / week (1 hour) for 10 weeks leading towards the second step of 1 skill session / week for 1 hour under instructor supervision for 6 weeks.
  Arms: Conventional method of Palliative care Training (Group A)
Other: Pedagogical (LWPPR) method of Palliative care Training (Group B) — Group B will receive training through the 5-steps pedagogy method including: the 1st step (learn), in which didactic lectures will be given to the students leading to the 2nd step (video watch), a 30 minutes video on Palliative care. The students first see the video in the class on multimedia with explanation and then share to the students in what's up group for frequent watching as per need. In the 3rd step (practice), students practiced their skills on a low fidelity simulator under instructor supervision on a scheduled day of the week in the nursing skill lab for 6 weeks. The errors will be corrected on the spot. A total of 11 groups will make with a ratio of 5 in each group. In the 4th step (perform), students perform their skill in real-life situations through the clinical rotation under supervision. Finally, the 5th step (Retain) will be established through self-directed learning in which an additional one-hour skill session / week will be provided to the students.
  Arms: Pedagogical (LWPPR) method of Palliative care Training (Group B)

SUMMARY:
Palliative care is a complex concept in nursing that needs special education and training. However, it is not focused and under-recognized discipline and the same is consistent with nursing students. In Pakistan, conventional teaching methods in nursing have been dominating all over. These methods are insufficient to meet the evolving needs of palliative care education. Hence, it is vital to explore new innovate approaches for palliative care education. Therefore, the goal of this clinical trial is to test a palliative care training program and its impact on experiential learning among senior student Nurses. The study compares the palliative care training through 5 step pedagogical method versus traditional method. Researchers will compare palliative care training program through 5-step pedagogical framework to 2-step conventional method to see is 5-step pedagogical framework is more effective in enhancing experiential learning in palliative care among senior nursing students compare to conventional method. The group 1 receives palliative care education through 2-step method in which didactic lecture and Simulation session provided. The group 2 receive palliative care education through a 5-step pedagogy in which expose to lecture, Simulation session, video, clinical and self-directed learning session. After intervention the experiential learning will be assessed based on knowledge, skill, and self-efficacy questionnaire.

DETAILED DESCRIPTION:
The nursing education often lack or little exposure to palliative care in undergraduate studies. In Pakistan, conventional teaching methods in Nursing have been dominating all over. In which students have little or no exposure of dying patients in clinical setting. Therefore, it is vital to explore new innovate approaches for palliative care education. The skill of nursing students influenced either positive or negative due to their educational method during training. In Pakistan conventional methods are dominant in nursing education. However, conventional methods are inadequate to impart practical knowledge among students. Previously, many studies reported interactive methods are dominant over the traditional methods to enhance competency and eventually employment opportunities. Hence, the ultimate goal of this study will be to see the effectiveness of palliative care training program among senior student nurses and its impact in experiential learning in nursing education. That will give the student nurses an opportunity to augment their proficiencies and improve knowledge in an innocuous environment. Eventually, the study will describe the strategies for effective learning and its impact on experiential leaning in nursing education.

This study will investigate the effectiveness of palliative care training and its impact on senior nursing student's experiential learning. The study will compare training through two different approaches a 2-step traditional approach and a 5-step pedagogy method and its impact on experiential learning. The experiential learning will be measured through the knowledge, competency and self-efficacy in palliative care as pre and post intervention using a single blind randomized controlled trial. The study may contribute in providing evidence of the efficacy of palliative care training in a resource limited setting. The study will contribute essentially in nursing education by investigating two different approaches and their effect on experiential learning.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students of 3rd and 4th year enrolled in the Bachelor of Science in Nursing for the academic year of 2025-2026
* Willing to attend the full course of palliative education.
* Have age of 18- 25 years.
* Both male and female will be included in the study.
* Those willing to give informed consent.

Exclusion Criteria:

* Will be on leave during study period

  * Have already received any educational training on palliative care.
  * Working as nursing assistants in any palliative care setting.
  * Have supply in the previous academic year.
  * Have previous exposure of working in palliative or end of life care services.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge Questionnaire | after 6 weeks of intervention and 3 months after intervention
  1. Knowledge: is considering awareness regarding palliative care. It will be measured through a 20-item true, false, and I don't know item scale called the Palliative Care Quiz for Nursing (PCQN), that measure palliative care knowledge among nursing students. The total score ranged from 0 to 20 and will be graded for each student as poor, average and good
Self-Efficacy | after 6 weeks of intervention and 3 months after intervention
  Self-efficacy is the professed capability to manage common aspects of palliative care. It will be measured through a 12-item scale called the Palliative Care Self-Efficacy Scale (PCSES). The total score ranged from 0 to 48 and will be graded for each student as low, moderate and good
Competency | after 6 weeks of intervention and 3 months after intervention
  is the ability of undergraduate nurse's skill of providing palliative care in clinical practice. It will be measured through Creighton Competency Evaluation Instrument in palliative care (CCEI-PC) in four areas of 1) assessment, 2) communication, 3) clinical judgment, and 4) patient safety. The total score ranged from 0-23 and will be graded as poor, average and good

CONTACTS AND LOCATIONS:
Overall Officials: Mishal Liaqat, PhD Scholar, Principal Investigator — Lincoln University College, Malysia; Dr. Regidor III Poblete Dioso, Study Chair — Lincoln University College, Malysia
Locations (2):
- Pakistan (2):
  - Al-Aleem Institute of Nursing, Gulab Devi Educational complex, Lahore, Lahore, Punjab Province
  - Rai Foundation College of Nursing, Sargodha, Punjab Province

IPD SHARING:
Plan to Share IPD: No